CLINICAL TRIAL: NCT02407028
Title: Hyperbaric Oxygen Brain Injury Treatment (HOBIT) Trial
Brief Title: Hyperbaric Oxygen Brain Injury Treatment Trial
Acronym: HOBIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gaylan Rockswold (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Strategies to Innovate EmeRgENcy Care Clinical Trials Network (Network)
Responsible Party: Sponsor-Investigator, Gaylan Rockswold, M.D., Neurosurgery, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: GLR-NIH-2015
Record Dates: First submitted 2015-03-18; First posted 2015-04-02 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Hyperbaric oxygen (1.5 ATA, no NBH) (Experimental): Hyperbaric oxygen at 1.5 ATA for 1 hour without NBH. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (1.5 ATA, no NBH)
- Hyperbaric oxygen (2.0 ATA, no NBH) (Experimental): Hyperbaric oxygen at 2.0 ATA for 1 hour without NBH. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (2.0 ATA, no NBH)
- Hyperbaric oxygen (2.5 ATA, no NBH) (Experimental): Hyperbaric oxygen at 2.5 ATA for 1 hour, without NBH. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (2.5 ATA, no NBH)
- Hyperbaric oxygen (1.5 ATA + NBH) (Experimental): Hyperbaric oxygen at 1.5 ATA for 1 hour and NBH for 3 hours. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (1.5 ATA + NBH)
- Hyperbaric oxygen (2.0 ATA + NBH) (Experimental): Hyperbaric oxygen at 2.0 ATA for 1 hour and NBH for 3 hours. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (2.0 ATA + NBH)
- Hyperbaric oxygen (2.5 ATA + NBH) (Experimental): Hyperbaric oxygen at 2.5 ATA for 1 hour and NBH for 3 hours. This treatment is administered twice a day for 5 days.
  Interventions: Drug: Hyperbaric oxygen (2.5 ATA + NBH)
- Normobaric Hyperoxia (NBH) (Experimental): Normobaric Hyperoxia (NBH meaning 100% O2 at 1.0 ATA) for 4.5 hours twice a day for 5 days.
  Interventions: Drug: Normobaric Hyperoxia (NBH)
- Usual care (Active Comparator): Usual care for severe TBI
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Hyperbaric oxygen (1.5 ATA, no NBH) — HBO at 1.5 ATA for 60 minutes without NBH. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (1.5 ATA, no NBH)
Drug: Hyperbaric oxygen (2.0 ATA, no NBH) — HBO at 2.0 ATA for 60 minutes without NBH. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (2.0 ATA, no NBH)
Drug: Hyperbaric oxygen (2.5 ATA, no NBH) — HBO at 2.5 ATA for 60 minutes without NBH. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (2.5 ATA, no NBH)
Drug: Hyperbaric oxygen (1.5 ATA + NBH) — HBO at 1.5 ATA for 60 minutes followed by NBH for 3 hours. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (1.5 ATA + NBH)
Drug: Hyperbaric oxygen (2.0 ATA + NBH) — HBO at 2.0 ATA for 60 minutes followed by NBH for 3 hours. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (2.0 ATA + NBH)
Drug: Hyperbaric oxygen (2.5 ATA + NBH) — HBO at 2.5 ATA for 60 minutes followed by NBH for 3 hours. Treatment will be twice a day for five days or until patient is following commands or brain dead
  Other Names: HBO
  Arms: Hyperbaric oxygen (2.5 ATA + NBH)
Drug: Normobaric Hyperoxia (NBH) — 100% fraction of inspired oxygen (FiO2) for 4.5 hours twice a day for five days or until patient following commands or brain dead
  Other Names: NBH
  Arms: Normobaric Hyperoxia (NBH)
Other: Usual Care — Will be treated with usual and customary care for severe traumatic brain injury
  Other Names: Standard of Care
  Arms: Usual care

SUMMARY:
The purpose of this innovative adaptive phase II trial design is to determine the optimal combination of hyperbaric oxygen treatment parameters that is most likely to demonstrate improvement in the outcome of severe TBI patients in a subsequent phase III trial.

DETAILED DESCRIPTION:
Preclinical and clinical investigations strongly indicate that hyperbaric oxygen (HBO2) is physiologically active in improving the destructive processes in severe Traumatic Brain Injury (TBI). However, prior to a definitive efficacy study, important information is required regarding optimizing the HBO2 treatment paradigm instituted in terms of pressure and whether NBH enhances the clinical effectiveness of the HBO2 treatment. Preclinical investigators working with TBI models have used pressures varying from 1.5 to 3.0 atmospheres absolute (ATA). Clinical investigators have used pressure varying from 1.5 to 2.5 ATA. However, the lungs in severe TBI patients have frequently been compromised by direct lung injury and/or acquired ventilator pneumonia and are susceptible to oxygen (O2) toxicity. Working within these constraints, it is essential to determine the most effective HBO2 treatment parameters without producing O2 toxicity and clinical complications. This proposed clinical trial is designed to answer these questions and to provide important data to plan a definitive efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older and 65 years or younger
* Present with severe TBI, defined as Glasgow Coma Scale (GCS) of 3 to 8.
* Marshall computerized tomography (CT) score >1 in patients with a GCS of 7 or 8 or patients with an alcohol level >200 mg/dl
* Ability to initiate the first hyperbaric oxygen treatment within 8 hours of admission in patients not requiring a craniotomy/craniectomy or any other major surgical procedure OR
* Ability to initiate the first hyperbaric oxygen treatment within 14 hours of admission in patients requiring a craniotomy/craniectomy or major surgical procedure

Exclusion Criteria:

* First hyperbaric oxygen treatment cannot be initiated within 24 hours of injury
* GCS of 3 with mid-position and non-reactive pupils bilaterally (4mm)
* Penetrating head injury
* Pregnant
* Pre-existing neurologic disease (e.g. TBI or stroke or neurodegenerative disorder) with confounding residual neurologic deficits
* Unstable acute spinal cord injury
* Fixed coagulopathy
* Severe hypoxia
* Cardiopulmonary resuscitation performed
* Coma suspected to de due to primarily non-TBI causes
* Any contraindications to the study intervention

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2028-10-26 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOS-E) | Assessment at 6 months

SECONDARY OUTCOMES:
Duration of ICP elevation | First 5 days
  The duration of ICP elevation will be measured using the area under the curve methodology
Therapeutic intensity level scores for controlling intracranial pressure (ICP) | First 5 days
  This tracks the level of therapies used to control ICP during the first 5 days
Brain tissue partial pressure of oxygen | First 5 days
  This outcome will be measured only in patients with LICOX monitoring
Serious adverse events | 180 days
  Events resulting in death, a life-threatening adverse event, or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
Peak brain tissue oxygen (P02) during HBO treatments | First 5 days
  To examine the association between peak brain tissue PO2 during hyperbaric treatment and favorable outcome at 6-months (measured by the GOS-E).

CONTACTS AND LOCATIONS:
Overall Officials: Gaylan L Rockswold, M.D., Ph.D., Principal Investigator — Hennepin County Medical Center, Minneapolis; William Barsan, MD, Principal Investigator — University of Michigan; Byron Gajewski, Ph.D., Principal Investigator — University of Kansas Medical Center; Frederick K Korley, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (11):
- United States (10):
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - St. Mary's Medical Center, West Palm Beach, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Hennepin County Hospital, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- Hamilton Heath Services, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gajewski BJ, Meinzer C, Berry SM, Rockswold GL, Barsan WG, Korley FK, Martin RH. Bayesian hierarchical EMAX model for dose-response in early phase efficacy clinical trials. Stat Med. 2019 Jul 30;38(17):3123-3138. doi: 10.1002/sim.8167. Epub 2019 May 9. PMID 31070807
- [Background] Gajewski BJ, Berry SM, Barsan WG, Silbergleit R, Meurer WJ, Martin R, Rockswold GL. Hyperbaric oxygen brain injury treatment (HOBIT) trial: a multifactor design with response adaptive randomization and longitudinal modeling. Pharm Stat. 2016 Sep;15(5):396-404. doi: 10.1002/pst.1755. Epub 2016 Jun 15. PMID 27306921
- [Background] Rockswold SB, Rockswold GL, Zaun DA, Zhang X, Cerra CE, Bergman TA, Liu J. A prospective, randomized clinical trial to compare the effect of hyperbaric to normobaric hyperoxia on cerebral metabolism, intracranial pressure, and oxygen toxicity in severe traumatic brain injury. J Neurosurg. 2010 May;112(5):1080-94. doi: 10.3171/2009.7.JNS09363. PMID 19852540
- [Background] Rockswold SB, Rockswold GL, Zaun DA, Liu J. A prospective, randomized Phase II clinical trial to evaluate the effect of combined hyperbaric and normobaric hyperoxia on cerebral metabolism, intracranial pressure, oxygen toxicity, and clinical outcome in severe traumatic brain injury. J Neurosurg. 2013 Jun;118(6):1317-28. doi: 10.3171/2013.2.JNS121468. Epub 2013 Mar 19. PMID 23510092